CLINICAL TRIAL: NCT04497103
Title: Effect of Task Oriented Training and Xbox KinectTM on Hand Function in Pediatric Burn
Acronym: HandBurn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, Department of Physical Therapy, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah., Qassim University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2694PT
Record Dates: First submitted 2020-07-24; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Burns; Hand Burn
Keywords: children burns; Hand Function; Grip strength; pinch strength; Jebsen-Taylor Hand Function Test; Duruoz Hand Index; Canadian Occupational Performance Measure
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Task-oriented training TOT group and Xbox training group were conducted with an average of 50-min sessions three times a week for 8 weeks.
  The traditional rehabilitation program conducted for 40-min sessions, three times per week for 8 weeks for all children.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Active Comparator): The traditional rehabilitation program conducted for 40-min sessions, three times per week for 8 weeks for all children.
  Interventions: Other: control
- task oriented training (Experimental): Task-oriented training TOT group was conducted with an average of 50-min sessions three times a week for 8 weeks. Baseline Canadian Occupational Performance Measure COPM results were used to generate individualized intervention goals for each participant.
  Interventions: Other: control; Other: task oriented training
- Xbox kinect (Experimental): Xbox training group was conducted with an average of 50-min sessions three times a week for 8 weeks. Baseline Canadian Occupational Performance Measure COPM results were used to generate individualized intervention goals for each participant.
  Interventions: Other: control; Other: Xbox kinect

INTERVENTIONS:
Other: control — The traditional therapy included immersing the hand in paraffin for 10 min; soft massaging with a moisturizing gel for 5 min; passive mobilization of the wrist, MP, PIP, and DIP joints; active/passive ROM and stretching exercises; strengthening exercises (done in static mode initially and progressed in the second month to dynamic strengthening using elastic bands); desensitizing sensory stimulation of hypertrophic scars, occupational therapy.
Other: Xbox kinect — The traditional plus Xbox Kinect games were related to five target activities determined according to the person-centered analysis results were chosen for each patient.
  Arms: Xbox kinect
Other: task oriented training — The traditional plus the target activities involved training with the materials (clothes, spoons, pencils, buttons, rope, etc) needed for the activity as well as Velcro cylinders, skill cubes, exercise bands, screw sets, therapeutic putty, and tripled coordination tools.
  Arms: task oriented training

SUMMARY:
The Jebsen-Taylor Hand Function Test and Canadian Occupational Performance Measure (COPM) were considered as primary outcome measurements. Secondary outcomes included total active range of motion (ROM) of the digits, hand grip strength and pinch strengths (tip, palmer and lateral pinch). All measurement was conducted at two occasions: at the baseline and after intervention.

DETAILED DESCRIPTION:
The included participant were children with a deep partial thickness or a full thickness burn induced by either a scaled or a flame thermal burn with involvement of more than 50% of the hand and wrist, total body surface area (TBSA) less than 30% , age ranged from 7 to 14 years, recent discharge of inpatient acute care, spontaneous healing (within 34 weeks) or grafting with split thickness or full-thickness skin grafts (at least before 2 weeks). Children were excluded from this study if they had infection, juvenile arthritis, fracture, tendon injuries, muscle injury, degenerative joint diseases, peripheral nerve diseases, Pre - established psychologically and physically disorders (extreme aphasia, cognitive and developmental deficits that can influence the rehabilitation).

ELIGIBILITY:
Inclusion Criteria:

* children with deep partial thickness or a full thickness burn
* burn induced by either a scaled or a flame thermal burn
* involvement of more than 50% of the hand and wrist
* total body surface area (TBSA) less than 30%
* age ranged from 7 to 14 years
* recent discharge of inpatient acute care
* spontaneous healing (within 34 weeks)
* grafting with split thickness or full-thickness skin grafts (at least before 2 weeks).

Exclusion Criteria:

* children with infection
* juvenile arthritis
* fracture
* tendon injuries
* muscle injury
* degenerative joint diseases
* peripheral nerve diseases
* Pre - established psychologically and physically disorders
* extreme aphasia
* cognitive and developmental deficits that can influence the rehabilitation

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test | baseline
  is an objective and standard method designed to assess the hand's functional abilities
Jebsen-Taylor Hand Function Test | immediately after the intervention
  is an objective and standard method designed to assess the hand's functional abilities
Duruoz Hand Index | baseline
  is a self-reported questionnaire developed to assess hand ability in the kitchen, during dressing, while performing personal hygiene and office tasks, and other general items
Duruoz Hand Index | immediately after the intervention
  is a self-reported questionnaire developed to assess hand ability in the kitchen, during dressing, while performing personal hygiene and office tasks, and other general items
Canadian Occupational Performance Measure | baseline
  is a client centered, occupation-focused outcome measure for the detection of change in perceived occupational performance over time.
Canadian Occupational Performance Measure | immediately after the intervention
  is a client centered, occupation-focused outcome measure for the detection of change in perceived occupational performance over time.

SECONDARY OUTCOMES:
total active range of motion (ROM) of the digits | baseline
  The total active ROM was measured by a hand-held steel finger goniometer
total active range of motion (ROM) of the digits | immediately after the intervention
  The total active ROM was measured by a hand-held steel finger goniometer
hand grip strength | baseline
  Grip strength was assessed using a Jamar hydraulic dynamometer
hand grip strength | immediately after the intervention
  Grip strength was assessed using a Jamar hydraulic dynamometer
pinch strength | baseline
  pinch strengths (tip, palmer and lateral pinch) were assessed using a pinch dynamometer
pinch strength | immediately after the intervention
  pinch strengths (tip, palmer and lateral pinch) were assessed using a pinch dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Maged Basha, PhD, Principal Investigator — Qassim University
Locations (1):
- Shorook Physical Therapy Centers, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables,and figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication.
Access Criteria: IPD will be available upon reasonable request by email from the main author after revising the requester qualification relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Result] Parry I, Painting L, Bagley A, Kawada J, Molitor F, Sen S, Greenhalgh DG, Palmieri TL. A Pilot Prospective Randomized Control Trial Comparing Exercises Using Videogame Therapy to Standard Physical Therapy: 6 Months Follow-Up. J Burn Care Res. 2015 Sep-Oct;36(5):534-44. doi: 10.1097/BCR.0000000000000165. PMID 26335108
- [Result] Voon K, Silberstein I, Eranki A, Phillips M, Wood FM, Edgar DW. Xbox Kinect based rehabilitation as a feasible adjunct for minor upper limb burns rehabilitation: A pilot RCT. Burns. 2016 Dec;42(8):1797-1804. doi: 10.1016/j.burns.2016.06.007. Epub 2016 Jul 9. PMID 27402183
- [Derived] Kamel FAH, Basha MA. Effects of Virtual Reality and Task-Oriented Training on Hand Function and Activity Performance in Pediatric Hand Burns: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Jun;102(6):1059-1066. doi: 10.1016/j.apmr.2021.01.087. Epub 2021 Feb 20. PMID 33617863